CLINICAL TRIAL: NCT06857006
Title: UAB 2507 - Randomized Phase II Study of Differential Margins in Single Isocenter Radiosurgery of Brain Metastases
Brief Title: Trial of Differential Margins in Single Isocenter Radiosurgery of Brain Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, John Fiveash, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300014291 (UAB2507); Robert Award (Other: The University of Alabama at Birmingham)
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Brain Metastases
Keywords: Brain Metastases; stereotactic radiosurgery (SRS); radiosurgery (RS); edge linear accelerator; single isocenter radiosurgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients will be blinded but the treating team will not be blinded after both plans are generated and clinically reviewed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0mm margin (Active Comparator): For each patient two radiation treatment plans will be created. One will have 0 mm margin for the planning target volume.
  Tumors will be prescribed based upon the maximum diameter of the largest tumor and location at the discretion of the treating radiation oncologist with the following guidance:
  < 2.0 cm diameter 16-20 Gy 2.0-4.0 cm diameter 3 fractions of 9 Gy for total 27 Gy.
  Interventions: Procedure: brain metastases radiosurgery
- 2mm margin (Active Comparator): For each patient two radiation treatment plans will be created. One will be 2 mm margin for the planning target volume.
  Tumors will be prescribed based upon the maximum diameter of the largest tumor and location at the discretion of the treating radiation oncologist with the following guidance:
  < 2.0 cm diameter 16-20 Gy 2.0-4.0 cm diameter 3 fractions of 9 Gy for total 27 Gy.
  Interventions: Procedure: brain metastases radiosurgery

INTERVENTIONS:
Procedure: brain metastases radiosurgery — Radiosurgery is the use of a focal high dose of radiation therapy to ablate or kill a tumor. This trial will enroll patients with brain metastases 4 cm or less in greatest diameter and will compare 0mm margin to a 2mm margin for treatment.

SUMMARY:
Radiosurgery is the use of a focal high dose of radiation therapy to ablate or kill a tumor. This trial will enroll patients with brain metastases 4 cm or less in greatest diameter and will compare 0mm margin to a 2mm margin for treatment.

DETAILED DESCRIPTION:
Without a stereotactic frame there is considerable variation in practice in the use of planning target volume (PTV) margins for linac radiosurgery. In particular, the use of a single isocenter for multiple targets geometrically increases the risk that rotational errors will result in significant dosimetric errors, and many centers have considered adding margin. A recent AAPM task group survey has found that ~90% of centers worldwide add a PTV margin to account for error and that 8% add more than 2 mm. The most common margin is 2 mm. Other potential reasons to add a margin include spacial MRI error, couch walkout, CBCT to linac isocenter mismatch, and undetected intrafraction motion. Treatment volume is the greatest predictor of radiation toxicity associated with radiosurgery and potentially unnecessary margins will lead to increased risk to the patient. This trial will incorporate a composite endpoint that includes control of the tumor and toxicity.

Uncomplicated tumor control probability (UTCP) is defined as the chance the tumor is locally controlled (TCP) without grade 3 or greater CNS toxicity (1-NTCP). The investigators hypothesize a 2 mm margin will worsen uncomplicated control compared to a 0 mm PTV margin in the treatment multiple metastases in a single fraction.

This trial will inform the standard of care margin (0 mm vs 2 mm) for single isocenter treatment of multiple targets.

ELIGIBILITY:
Inclusion Criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male or female, aged 19 and older
3. Brain metastases diagnosis not requiring retreatment to the same tumor
4. For females of reproductive potential should undergo pregnancy testing as per UAB Radiation Oncology standard policies
5. Ability of subject or Legally Authorized Representative (LAR)) to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Current use of cytotoxic chemotherapy within 3 days of treatment. There are no restrictions on the use of immunotherapy during treatment. TKIs known to be radiation sensitizers such as BRAF should be held at least 24 hours prior to treatment.
2. Inability to have MRI imaging
3. Pregnancy
4. Treatment with another investigational drug 14 days of enrollment
5. Radiosurgery planned for post-operative adjuvant cavity only. Patients with any gross residual after surgery are eligible. Patients with at least one intact metastasis may enroll but adjuvant cavity will not be evaluable.
6. At the time of Radiation Oncology consultation more than twenty targets are identified. Note that it is common that a few additional metastases may be identified during the treatment planning or peer review processes. More than twenty targets may be included if this number is found after the initial clinical review of the treatment planning MRI.
7. Tumor maximal diameter > 4 cm.
8. Prior SBRT or SRS to a lesion planned for retreatment. Note that patients with prior whole brain radiation alone are eligible.
9. Patients with diffuse leptomeningeal tumor are not eligible. Patients with a focal dural or pachymeningeal tumor are eligible if other intra-axial tumors are planned to be treated. Similar to postoperative cavities, the pachymeningeal tumor deposit will be treated but not evaluable for the assessment of local control or toxicity.

INCLUSION OF VULNERABLE PARTICIPANTS Vulnerable populations as defined by the NIH including children, prisoners, and adult subjects who lack capacity to consent to research participation are not eligible.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Difference between 0mm and 2mm | 12 months
  Fisher's Exact Test to determine if (per patient) uncomplicated control is improved or worsened with the addition of a 2mm PTV margin in the treatment of brain metastases with single isocenter radiosurgery.

SECONDARY OUTCOMES:
Maximum margin size of the tumor | 12 months
  To compare 0mm margin and 2mm margin radiosurgery for local tumor control, RANO assessment by individual tumor calculated by multiplying the longest diameter on an axial slice and its longest perpendicular diameter on the same slice
Percentage of toxicity | 12 months
  To compare 0mm margin and 2mm margin radiosurgery for toxicity. NTCP - assessed per tumor and per patient, assign to all tumors if attribution ambiguous (only grade 3 or greater CNS toxicity included)
Change in normal brain dosimetry | 12 months
  To compare 0mm margin and 2mm margin radiosurgery for normal brain dosimetry.
  * Dosimetry of normal brain (2 mm vs 0 mm)
  * Dosimetry of hippocampi (2 mm vs 0 mm)

CONTACTS AND LOCATIONS:
Overall Officials: John A Fiveash, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham (UAB) Hazelrig-Salter Radiation Oncology Center, Birmingham, Alabama, United States